CLINICAL TRIAL: NCT04661085
Title: A Descriptive Study of Patients Suspected With Infection in the Emergency Department, With a Special Focus on Infection With Unknown Origin.
Brief Title: Infection With Unknown Origin in the Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-ED-11f-2020
Record Dates: First submitted 2020-12-08; First posted 2020-12-09 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Infection
Keywords: antibiotics; source; diagnosis; fever; pyrexia
MeSH Terms: conditions — Infections; Disease; Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a suspected infection: Acutely admitted patients from the emergency department across 3 sites who have a suspected infection.
  Interventions: Diagnostic Test: Broader Medical history and clinical tests

INTERVENTIONS:
Diagnostic Test: Broader Medical history and clinical tests — Patients will be treated with standard care plus additional blood tests, urine culture and urine flow cytometry,

SUMMARY:
Patients suspected with infection is one of the major groups, who are admitted to the Danish Emergency Departments (ED). Currently, there is no overall description of the distribution of these infections. The aim of this study is to characterize ED patients with a suspected infection whereby the focus of the infection is of an unknown origin.

DETAILED DESCRIPTION:
Bacteria resistant to antibiotics are associated with high antibiotic consumption and are identified by the World Health Organisation as a major public health threat. Despite efforts to optimize antibiotic consumption in Denmark, the total consumption in the hospital sector increased from 2009-2018 and the incidence of multi-resistance bacteria (MRB) is increasing. A Danish multicenter study has shown that every 20th patient in the emergency department has MRB. Patients with an infection of unknown origin tend to be prescribed a broad-spectrum antibiotic, as physicians endeavour to target probable origins in the body. The uncertainty associated with the diagnosis may lead to an overconsumption of antibiotics, which contributes to increased development of resistant bacteria and threatens future treatment options.

The aim of this study is to characterize patients admitted to the ED suspected with infection. The study will have three objectives:

* To describe the distribution of ED infections according to the registered diagnosis in the medical record compared to a clinical expert panel assessment
* To identify clinically relevant information available at admission associated with a patients infection of unknown origin.
* To investigate the association between an adverse event and clinically relevant information for patients with infection of unknown origin

The investigators' hypothesis is that with an improvement of knowledge about patients with an infection of unknown origin, a more accurate diagnosis can be made leading to a more appropriate antibiotic therapy and contributing to the fight against resistance to antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Adults admitted to the ED will be invited to participate in the study, if the physician, receiving the patient, suspect the patient has an infection (e.g. indication for blood culture).

Exclusion Criteria:

* If the attending physician considers that participation will delay a life-saving treatment or patient needs direct transfer to the intensive care unit.
* Admission within the last 14 days
* Verified COVID-19 disease within 14 days before admission
* Pregnant women
* Severe immunodeficiencies: Primary immunodeficiencies and secondary immunodeficiencies (HIV positive CD4 <200, Patients receiving immunosuppressive treatment (ATC L04A), Corticosteroid treatment (>20 mg/day prednisone or equivalent for >14 days within the last 30 days), Chemotherapy within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acutely admitted patients suspected with infection at three hospitals in the region of Southern Denmark - Hosptial Sonderjylland, Hospital Lillebaelt and Odense University Hospital.
Sampling Method: Probability Sample
Enrollment: 966 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis after 2 days | 48 hours after admission emergency department
  Diagnosis code of patient (registered medical record and clinical expert panel assessment)

SECONDARY OUTCOMES:
Intensive care unit treatment | within 60 days from admission to the emergency department
  Transfer to the intensive care unit will be recorded during the current hospitalization as a binary variable (transferred/not-transferred)
Length of stay | within 60 days from admission to the emergency department
  Defined as the time (in days) spent in hospital during the current admission. Measured in days from admission to hospital discharge. Discharge date minus admission date
30-days mortality | within 30 days from admission to the emergency department
  Mortality within 30 days from admission to the Emergency Department
Readmission | within 30 days from day of discharge
  Binary
In-hospital mortality | within 60 days from admission to the emergency department
  binary
Diagnose code at hospital discharge | within 60 days from admission to the emergency department
  code registered in medical record at discharge

OTHER OUTCOMES:
90-day mortality | Within 90 days from admission to emergency department
  Mortality - binary
Level of infection markers | Within 4 hours of arrival to emergency department
  concentration of serum procalcitonin, CRP and suPAR
Level of markers of lung injury | Within 4 hours of arrival to emergency department
  concentration of serum surfactant protein D, KL-6, and YKL-40
Bacteriuria | Within 4 hours of arrival to emergency department
  defined by microbiologist on urine culture analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, Study Chair — University Hospital of Southern Denmark
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carter-Storch R, Olsen UF, Mogensen CB. Admissions to emergency department may be classified into specific complaint categories. Dan Med J. 2014 Mar;61(3):A4802. PMID 24814917
- [Background] Bager F. DANMAP: monitoring antimicrobial resistance in Denmark. Int J Antimicrob Agents. 2000 May;14(4):271-4. doi: 10.1016/s0924-8579(00)00135-7. PMID 10794946
- [Background] Skjot-Arkil H, Mogensen CB, Lassen AT, Johansen IS, Chen M, Petersen P, Andersen KV, Ellermann-Eriksen S, Moller JM, Ludwig M, Fuglsang-Damgaard D, Nielsen FE, Petersen DB, Jensen US, Rosenvinge FS. Carrier prevalence and risk factors for colonisation of multiresistant bacteria in Danish emergency departments: a cross-sectional survey. BMJ Open. 2019 Jun 27;9(6):e029000. doi: 10.1136/bmjopen-2019-029000. PMID 31253624
- [Background] Zhao MZ, Ruan QR, Xing MY, Wei S, Xu D, Wu ZH, Zhu L, Zhu JL, Zheng CF, Liu S, Yu ZJ, Qi JY, Song JX. A Diagnostic Tool for Identification of Etiologies of Fever of Unknown Origin in Adult Patients. Curr Med Sci. 2019 Aug;39(4):589-596. doi: 10.1007/s11596-019-2078-3. Epub 2019 Jul 25. PMID 31346995
- [Background] Courjon J, Demonchy E, Degand N, Risso K, Ruimy R, Roger PM. Patients with community-acquired bacteremia of unknown origin: clinical characteristics and usefulness of microbiological results for therapeutic issues: a single-center cohort study. Ann Clin Microbiol Antimicrob. 2017 May 19;16(1):40. doi: 10.1186/s12941-017-0214-0. PMID 28526094
- [Derived] Skjot-Arkil H, Cartuliares MB, Heltborg A, Lorentzen MH, Hertz MA, Kaldan F, Specht JJ, Graumann O, Lindberg MJH, Mikkelsen PA, Nielsen SL, Jensen J, Roge BT, Rosenvinge FS, Mogensen CB. Clinical characteristics and diagnostic accuracy of preliminary diagnoses in adults with infections in Danish emergency departments: a multicentre combined cross-sectional and diagnostic study. BMJ Open. 2024 Dec 5;14(12):e090259. doi: 10.1136/bmjopen-2024-090259. PMID 39638587
- [Derived] Skjot-Arkil H, Heltborg A, Lorentzen MH, Cartuliares MB, Hertz MA, Graumann O, Rosenvinge FS, Petersen ERB, Ostergaard C, Laursen CB, Skovsted TA, Posth S, Chen M, Mogensen CB. Improved diagnostics of infectious diseases in emergency departments: a protocol of a multifaceted multicentre diagnostic study. BMJ Open. 2021 Sep 30;11(9):e049606. doi: 10.1136/bmjopen-2021-049606. PMID 34593497